CLINICAL TRIAL: NCT07317544
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of ABS-201 in Healthy Adult Participants With and Without Androgenetic Alopecia
Brief Title: Study of ABS-201 Evaluating Single and Multiple Ascending Doses in Healthy Adults With and Without Androgenetic Alopecia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Absci Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABS-201-101
Record Dates: First submitted 2025-11-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Androgenetic Alopecia (AGA); Healthy Volunteers - Male and Female
Keywords: Androgenetic Alopecia; Hair Loss; AGA; Female hair loss; Male pattern baldness; hair regrowth
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Approximately 4-6 SAD IV doses will be tested and if safe and well tolerated, approximately 3-4 Sub-cutaneous MAD doses will be tested in participants with or without AGA.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- SAD IV Dose 1 - 150mg ABS201 or Placebo (Experimental): ABS-201 IV Single Dose
  Interventions: Drug: ABS-201 IV Single Dose; Drug: Placebo IV
- SAD IV Dose 2 - 450mg ABS201 or Placebo (Experimental): Single Intra-venous dose of active study drug or placebo in Healthy Volunteers
  Interventions: Drug: ABS-201 IV Single Dose; Drug: Placebo IV
- SAD IV Dose 3 - 900mg ABS201 or Placebo (Experimental): Single Intra-venous dose of active study drug or placebo in Healthy Volunteers
  Interventions: Drug: ABS-201 IV Single Dose; Drug: Placebo IV
- SAD IV Dose 4 - 1800mg ABS201 or Placebo (Experimental): Single Intra-venous dose of active study drug or placebo in Healthy Volunteers
  Interventions: Drug: ABS-201 IV Single Dose; Drug: Placebo IV
- MAD SC Dose 1 - 300mg ABS201 or Placebo (Experimental): Multiple Ascending Doses of active study drug or placebo delivered subcutaneously in Patients with AGA
  Interventions: Drug: ABS-201 SC Multiple Doses; Drug: Placebo SC Injection
- MAD SC Dose 2 - 600mg ABS201 or Placebo (Experimental): Multiple Ascending Doses of active study drug or placebo delivered subcutaneously in Patients with AGA
  Interventions: Drug: ABS-201 SC Multiple Doses; Drug: Placebo SC Injection
- MAD SC Dose 2 - 1200mg ABS201 or Placebo (Experimental): Multiple Ascending Doses of active study drug or placebo delivered subcutaneously in Patients with AGA
  Interventions: Drug: ABS-201 SC Multiple Doses; Drug: Placebo SC Injection

INTERVENTIONS:
Drug: ABS-201 IV Single Dose — ABS-201 is an IgG1 monoclonal antibody developed to specifically target the prolactin receptor (PRLR),
  Arms: SAD IV Dose 1 - 150mg ABS201 or Placebo; SAD IV Dose 2 - 450mg ABS201 or Placebo; SAD IV Dose 3 - 900mg ABS201 or Placebo; SAD IV Dose 4 - 1800mg ABS201 or Placebo
Drug: Placebo IV — Matching placebo
  Arms: SAD IV Dose 1 - 150mg ABS201 or Placebo; SAD IV Dose 2 - 450mg ABS201 or Placebo; SAD IV Dose 3 - 900mg ABS201 or Placebo; SAD IV Dose 4 - 1800mg ABS201 or Placebo
Drug: ABS-201 SC Multiple Doses — Multiple doses of ABS-201 for Subcutaneous injection
  Arms: MAD SC Dose 1 - 300mg ABS201 or Placebo; MAD SC Dose 2 - 1200mg ABS201 or Placebo; MAD SC Dose 2 - 600mg ABS201 or Placebo
Drug: Placebo SC Injection — Subcutaneous Placebo injection for MAD arms
  Arms: MAD SC Dose 1 - 300mg ABS201 or Placebo; MAD SC Dose 2 - 1200mg ABS201 or Placebo; MAD SC Dose 2 - 600mg ABS201 or Placebo

SUMMARY:
The goal of this clinical trial is to learn if ABS-201 (a new medication) is safe and tolerable when used to improve hair growth in men and women. The trial will start with healthy volunteers and if safe, will treat participants with certain types of hair loss.

The main questions it aims to answer are:

What medical problems, if any, do participants experience when taking a single dose or many doses of ABS-201? How does the medication, ABS-201, compare to placebo (a look alike substance that does not contain any medication).

Participants who qualify for the trial will receive either ABS-201 or a placebo, and visit the study clinic for scheduled checkups and tests for approximately 1 year.

ELIGIBILITY:
Inclusion Criteria (Major):

* Participants must be overtly healthy, as determined by medical evaluation, which includes a review of medical and surgical history, physical examination, and a 12-lead ECG.
* Must have normal ranges for hematology, clinical chemistry, coagulation tests, and urine analysis parameters
* Must have a body mass index (BMI) of 18 to 32 kg/m2, inclusive, at screening, with a total body weight >60 kg.
* Participants, male and female, must be willing to avoid pregnancy for the duration of the trial.
* Participants must be capable of giving signed informed consent
* Participants must have no signs or symptoms of active or latent tuberculosis (TB),

Additional Inclusion criteria for patients with AGA:

* Diagnosis of AGA with a Norwood-Hamilton Scale III vertex to V pattern.
* Willing to clip target hair area for analysis and avoid scalp pigmentation products.
* Willingness to maintain approximately the same hair length at each study visit
* Additional Inclusion Criteria for postmenopausal women with AGA: Diagnosis of AGA with a Ludwig Scale I-3, I-4, II-1, II-2 pattern, with a documented history of AGA for ≥12 months and no rapid progression (e.g., sudden shedding, acute diffuse thinning, or scarring alopecia) in the 6 months prior to screening.

Exclusion Criteria (Major):

* History or presence of cancer, except for basal cell carcinoma or cervical dysplasia successfully treated with no recurrence for ≥90 days before screening.
* History of liver disease, Gilbert's syndrome, or abnormal liver function tests (e.g., ALT, AST, or bilirubin > ULN) at screening
* Systolic blood pressure ≤90 or ≥140 mmHg, diastolic BP ≤40 or ≥90 mmHg, pulse rate <40 or >100 bpm
* Positive test for HIV, hepatitis B (HBV), or hepatitis C (HCV).
* Recent blood donation
* Any clinically significant psychiatric disorder
* Pregnant or breastfeeding females or those planning pregnancy during the study.
* History of postpartum depression, perimenopausal mood instability, or estrogen withdrawal syndrome

Additional Exclusion criteria for participants with AGA undergoing hair assessments:

* Prior use of hair loss treatments:

  1. Topical minoxidil within 3 months before screening.
  2. Oral minoxidil other hair growth stimulators within 6 months before screening.
  3. Finasteride within 6 months before screening
  4. Dutasteride within 12 months before screening.
* Use of GLP-1 receptor agonists (e.g., semaglutide, liraglutide, dulaglutide, exenatide, tirzepatide, or similar agents) within 3 months prior to screening
* History of hair transplantation or other major scalp procedures or planned procedures during the study.
* Use of hair extensions, wigs, hairpieces, weaves, or any other artificial hair enhancement methods within 30 days prior to screening and throughout the study.
* History of clinically significant dermatologic disease of the scalp that could interfere with hair assessments or target area imaging

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological males and biological females
Enrollment: 227 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of treatment-related adverse events | From enrollment to the end of the Study (SAD approximately 12 months, MAD approximately 18 months)
  Safety assessments based on reporting of Treatment Emergent Adverse Events

SECONDARY OUTCOMES:
CMAX | From enrollment to the end of the Study (SAD up to 12 months, MAD up to 18 months)
  Peak concentration: The highest blood concentration after study drug administration
AUC | From enrollment to the end of the Study (SAD up to 12 months, MAD up to 18 months)
  Area under the drug time curve: The area surrounded by the blood concentration curve to the time axis.
TMAX | From enrollment to the end of the Study (SAD up to 12 months, MAD up to 18 months)
  Peak time: The time required to reach peak concentration after study drug administration
Terminal elimination rate | Enrollment up to the End of Study (SAD up to 12 months, MAD up to 18 months)
  The terminal elimination rate constant is obtained from the linear regression of the phase elimination concentration point
Terminal elimination Half-life | From enrollment to the end of the Study (SAD up to 12 months, MAD up to 18 months)
  The time required for the terminal phase blood concentration to decrease by half
Change from Baseline in Prolactin | Enrollment up to End of Study (SAD up to 12 months, MAD up to 18 months)
  Change from baseline in PRL levels,
Change from Baseline in DHEA-S | Enrollment up to End of Study (SAD 12months or MAD 18 months)
  Change from baseline in dehydroepiandrosterone (DHEA-S)
Change from Baseline in IGF-1 | Enrollment up to the end of study (SAD 12 months or MAD 18 months)
  Change from Baseline in Insulin Growth Factor
Treatment Emergent Incidence of ADA | Enrollment up to End of Study (SAD 12 months or MAD 18 months)
  Measuring Incidence of Anti-Drug Affects (ADAs)
Treatment Emergent Incidence of NAb | Enrollment up to the End of Study (SAD 12 months, MAD 18 months)
  Measure the treatment emergent incidence of Neutralizing Antibodies (NAbs) in participants who have developed ADAs

OTHER OUTCOMES:
Change from Baseline in Total Area Hair Count (TAHC) | Enrollment and up to End of Study Visit (SAD 12 months, MAD 18 months)
  Measures the change from baseline in Total Area Hair Count (TAHC) in healthy adult participants with AGA.
Change from Baseline in Total Area Hair Width (TAHW) | Enrollment to the End of Study (SAD 12 months, MAD 18 months)
  Change from baseline in Total Area Hair Width (TAHW) in healthy adult participants with AGA.
Change From baseline Participant Self Assessment of Hair Growth | Enrollment up to End of Study (SAD 12 months, MAD 18 months)
  Hair Growth Assessment in participants with AGA using central photography images comparing baseline to later visits using a Subject Self-Assessment Scale. This scale is an ordinal scale with 7 options (Very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse). Improved scores suggest improved hair growth.
Change From baseline Investigator Global Assessment of Hair Growth | Enrollment to End of Study (SAD 12 months, MAD 18 months)
  Change from baseline in central photography images comparing baseline to later visits using an Investigator Global Assessment Scale. This scale is an ordinal scale with 7 options (Very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse). Improved scores suggest improved hair growth.
Change from Baseline in Target Area Hair Darkness/Pigmentation (TAHD) by Central Analysis of Macrophotography | Enrollment to End of Study (SAD 12 Months, MAD 18 Months)
  Change from baseline in TAHD is calculated using a Central Imaging analysis procedure for quantitatively measuring hair shafts. For each detected and segmented hair shaft, the average darkness is determined by calculating the darkness value of every pixel and then computing the mean. Darkness values range from 0 to 255, where 0 represents the darkest possible value and 255 represents the lightest.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Sinclair Dermatology, Melbourne, Victoria
  - Nucleus Network, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
The IPD sharing plan is not yet developed. The study team will consider data sharing at a later date.